CLINICAL TRIAL: NCT06727383
Title: Production and Expansion of Chimeric Antigen Receptor (CAR)-Natural Killer (NK) Cells From Patients Affected by Lympho or Myeloproliferative Disorders and From Healthy Donors
Brief Title: CAR-NK Cells Production and Expansion From Patients With Lympho or Myeloproliferative Disorders and From Healthy Donors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IEO 1886
Record Dates: First submitted 2024-03-19; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-03

CONDITIONS: Healthy Donors; Myeloproliferative Diseases; Lymphoproliferative Disorders
Keywords: CAR-NK cells; immunotherapeutic activity
MeSH Terms: conditions — Lymphoproliferative Disorders | interventions — Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort a (Experimental): The collection of PBMCs will be performed during standard blood test procedures: 40 mL of PB will be collected in 8 EDTA tubes.
  Interventions: Procedure: peripheral blood collection
- Cohort b (Experimental): The collection of CD34+ cells will be performed during HSC mobilization and staging bone marrow aspirations, as follows:
  1. During standard HSC mobilization, 10 mL peripheral blood will be collected in two EDTA tubes from patients with >20 CD34+ cells/mcL.
  2. 5 mL of bone marrow will be collected in one EDTA tube during bone marrow aspiration performed in the context of standard diagnostic procedures.
  Interventions: Procedure: peripheral blood collection
- Cohort c (Experimental): The collection of CD34+ cells will be performed from a LP required in the context of standard therapeutic procedures
  Interventions: Procedure: leukapheresis

INTERVENTIONS:
Procedure: peripheral blood collection — standard blood test procedures
  Arms: Cohort a; Cohort b
Procedure: leukapheresis — Leukapheresis is the procedure that allows the separation and collection of hematopoietic stem cells (HSCs) from peripheral blood. The collection takes place through a machine called a "cell separator": it uses centrifugal force to separate the mononuclear cells from all the other cells in the blood and plasma.
  Arms: Cohort c

SUMMARY:
Recent studies demonstrated the safety and efficacy of allogeneic and autologous infusion of NK cells as adoptive immunotherapy in malignant hematological diseases and solid tumors.NK cells are innate immunity effectors with antitumor activity regulated by a wide variety of receptors located on their cell surface, with both activating and inhibiting roles.Receptors with an inhibitory role include receptors of the KIRs family (Killer Immunoglobulin like Receptors) and receptors of the CD94 / NKG2A complex and are capable of recognizing molecules of Human Leukocyte Antigen class I (HLA-I). Receptors of the KIRs family are members of the immunoglobulin superfamily and are encoded by highly polymorphic genes located on chromosome 19q13.4 in a region known as a leukocyte receptor cluster (LCR). The predominant ligand for KIRs receptors is HLA-C, but other studies show that HLA-A and HLA-B are also involved. Receptors with an activating role, on the other hand, such as NCRs (Natural Cytotoxic receptors), are specific to NK cells, while other epitopes such as CD 56 are also present on other populations of T lymphocytes.

This receptor condition allows, in patients suffering from haemopathy and undergoing transplantation allogeneic stem cell, an alloreactivity induced by the mismatch between the donor's KIRs and their ligands on recipient target cells and, therefore, the role of NK cells as allogeneic effectors. The engraftment of NK cells has been shown to be correlated with a lower risk of disease recurrence, therefore the therapeutic infusion of NK cells from donors could allow, with benefit, the acquisition of fully functional NK cells in the recipient.

DETAILED DESCRIPTION:
The primary aim of the study is to manufacture and expand NK cells expressing CD19, CD79 and CD123 CARs from Peripheral Blood Mononucleated Cells (PBMCs) (cohort a) and from CD34+ cells (cohort b and c) of subjects affected by myelo or lymphoproliferative disorders or healthy donors.

The secondary aim is to evaluate their cytotoxic activity in preclinical models. The main steps of CAR-NK cell manufacturing and preparation are the followings

1. Collection of peripheral venous blood (40 mL collected in EDTA tubes for cohort a, or 10 mL from patients with >20 CD34+ cells/mcL for cohort b), or blood from bone marrow aspiration (5 mL of bone marrow collected in one EDTA tube for cohort b), or a part of LP (2 mL of PL in one EDTA tube for cohort c) from subjects with myelo/lymphoproliferative diseases and from Healthy Donors;
2. Selection of mononucleated cells through a density gradient centrifugation technique (Ficoll-Histopaque) (cohort a and b);
3. Selection of CD34 + Hematopoietic stem cells (HSCs) through magnetic activated cell sorting (cohort b)
4. Expansion NK cells from PBMCs (cohort a), using supplements such as recombinant cytokines, stimulatory antibodies, medicinal products and irradiated cells to support the process;
5. Expansion of CD34+ cells (cohort b and c), using supplements such as recombinant cytokines, stimulatory antibodies, medicinal products and irradiated cells to support the process, in order to promote differentiation to the NK cell lineage;
6. Engineering of NK cells through retroviral or lentiviral vectors (VL) that enable transduction with chimeric antigen receptors (CARs) specific for neoplastic cells.
7. Increasing the activation of NK cells through the down regulation of their inhibitory receptors (CRISPR Cas-9 technology and pharmacological modulation) or pharmacologic modulation of epigenetic, metabolic (HIF1-alpha) and immune-related pathways;
8. Testing, in in vitro and in vivo preclinical models, the persistence and the activity of the CAR-NK cells produced.

100 patients and 40 healthy donors will be prospectively enrolled over 3 years in order to perform 70 experiments of NK-cell expansion from PBMCs and 70 experiments from CD34+ cells (from PB or bone marrow or LP).

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 18 capable of understanding and willing
* Subjects affected by myelo/lymphoproliferative diseases

Exclusion Criteria:

* Patients with psychiatric, addictive, or any disorder, which compromises ability to give informed consent for participation in this study.
* Patients affected by lympho or myeloproliferative disorders and Healthy Donors with known acute and chronic viral and bacterial infections :HIV, HCV (Hepatitis C Virus), HBV (Hepatitis B Virus), syphilis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Primary objective | 3 years
  100 patients and 40 healthy donors will be prospectively enrolled over 3 years in order to perform 70 experiments of NK-cell expansion from PBMCs and 70 experiments from CD34+ cells (from PB or bone marrow or LP). We aim to demonstrate feasibility of the program (as defined in the primary endpoint) in 80% of eligible patients in the cohorts a), b) and c). The study will be powered to estimate the fraction of enrolled patients that obtain a full NK expansion defined as A) ≥40 fold ex-vivo expansion of the NK cell population at day 15 of cell culture and B) ≥1x10^9 NK-cells following ex-vivo expansion of 1x10^6 CD34+ cells at day 30 of cell culture; a minimum of 70 patients are required to estimate a true prevalence rate between 70 and 90% with 95% confidence interval (with 56 expected successful cases)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Derenzini, MD, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- Istituto Europeo di Oncologia, Milan, Italy

IPD SHARING:
Plan to Share IPD: No